CLINICAL TRIAL: NCT01771341
Title: Evaluation of Synchrony in the Post-operative Patient (NAVA vs Pressure Support)
Brief Title: Evaluation of Synchrony in the Post-operative Patient
Acronym: SYNCHRONY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2010.646
Record Dates: First submitted 2012-06-15; First posted 2013-01-18 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Patient-ventilator Asynchronism
Keywords: NAVA; post operative
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support (Placebo Comparator)
  Interventions: Device: MAQUET SERVOi ventilator
- NAVA (Experimental)
  Interventions: Device: MAQUET SERVOi ventilator with Edi Catheter

INTERVENTIONS:
Device: MAQUET SERVOi ventilator with Edi Catheter — NAVA respiratory modality
  Other Names: Neurally Adjusted Ventilatory Assist
  Arms: NAVA
Device: MAQUET SERVOi ventilator — Pressure Support
  Other Names: Pressure Support
  Arms: Pressure support

SUMMARY:
Neurally adjusted ventilatory support improved synchronization in the medical patient. However no data are available in the postoperative patient.

This way the investigators designed a prospective randomized cross over trial to evaluate this issue in the abdominal post-operative patient.

ELIGIBILITY:
Inclusion Criteria:

* adult > 18 yr-old
* abdominal post-operative patient
* able to trigger the ventilator

Exclusion Criteria:

* infant
* pregnancy
* esophageal surgery
* recent esophageal variceal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Asynchrony index (AI) | 8 hours
  Number of asynchrony events/total respiratory rate

SECONDARY OUTCOMES:
PaO2/FiO2 ratio | 8 hours
  ratio of partial pressure arterial oxygen and fraction of inspired oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Florent WALLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon- Centre Hospitalier Lyon Sud, Pierre-Bénite, France